CLINICAL TRIAL: NCT02194075
Title: Methylphenidate Hydrochloride Controlled-Release Tablets Augmentation Strategy for Patients With Obsessive Compulsive Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, sunnyrong, MD,PHD, Guangdong Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B2013006
Record Dates: First submitted 2014-07-11; First posted 2014-07-18 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2013-12

CONDITIONS: Obsessive Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fluvoxamine+Methylphenidate Hydrochloride (Active Comparator): Fluvoxamine: tablet, 100mg-300mg/d, were treated with a course of 8 weeks.
  Methylphenidate Hydrochloride: tablet, 18mg-36mg/d, were treated with a course of 8 weeks.
  Interventions: Drug: Fluvoxamine+Methylphenidate hydrochloride
- Fluvoxamine+sugar pill (Placebo Comparator): Fluvoxamine: tablet, 100mg-300mg/d, were treated with a course of 8 weeks.
  sugar pill: tablet, 1-2 tablets/d, were treated with a course of 8 weeks.
  Interventions: Drug: Fluvoxamine+sugar pill

INTERVENTIONS:
Drug: Fluvoxamine+Methylphenidate hydrochloride
  Arms: Fluvoxamine+Methylphenidate Hydrochloride
Drug: Fluvoxamine+sugar pill
  Arms: Fluvoxamine+sugar pill

SUMMARY:
Explore the efficacy of methylphenidate hydrochloride controlled-release tablets add-on pharmacotherapy on clinical symptomatology and cognitive functioning in a sample of patients with obsessive-compulsive disorder (OCD) receiving fluvoxamine maleate. To test the hypothesis that methylphenidate hydrochloride controlled-release tablets augmentation of fluvoxamine treatment is well tolerated and may be proposed as an effective therapeutic strategy to improve outcome in OCD.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Met DSM-V criteria
* Y-BOCS ≥ 16
* Course of illness ≥ 1year
* Age range between 18~40 years old
* Junior high school education level above

Exclusion Criteria:

* Any other psychiatric axis-I or axis-II disorders
* History of epileptic seizures or any other neurological disorder
* Any other clinically relevant abnormalities in their medical history or laboratory examinations; alcohol or drug abuser

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Yale-Brown Obsessive Compulsive Scale (Y-BOCS) | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong General Hospital, Guangdong academy of medical science, Guangzhou, Guangdong, China